CLINICAL TRIAL: NCT01245673
Title: Phase II Combination Immunotherapy After ASCT for Advanced Myeloma to Study MAGE-A3 Immunizations With Hiltonol® (Poly-ICLC) Plus Transfer of Vaccine-Primed Autologous T Cells Followed by Lenalidomide Maintenance
Brief Title: Combination Immunotherapy and Autologous Stem Cell Transplantation for Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 02710; UMGCC 0955 (Other: University of Maryland Greenebaum Cancer Center)
Record Dates: First submitted 2010-11-19; First posted 2010-11-22 (Estimated); Results first posted 2020-03-19 (Actual); Last update posted 2020-04-06 (Actual); Status verified 2020-03

CONDITIONS: Myeloma
Keywords: Advanced Disease; MAGE-A3 Immunizations with Hiltonol; Vaccine-Primed Autologous T-Cells; Lenalidomide Maintenance
MeSH Terms: conditions — Neoplasms, Plasma Cell | interventions — Heptavalent Pneumococcal Conjugate Vaccine; Lenalidomide; poly ICLC

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Prevnar, T Cells, Lenalidomide, MAGE A-3 (Experimental): All patients will receive a priming immunization with a MAGE-A3/GM-CSF vaccine with adjuvant Hiltonol® (Poly-ICLC) along with the pneumococcal conjugate vaccine/PCV control vaccine about 10 days before a steady-state mononuclear cell apheresis. Patients will then undergo hematopoietic stem cell mobilization. All patients will receive high-dose melphalan followed by hematopoietic stem cells on day 0. On day +2, patients will receive anti-CD3/anti-CD28-costimulated autologous T cells. At days 14, 42, and 90, patients will receive MAGEA3/GM-CSF (+Hiltonol® Poly-ICLC) and PCV booster immunizations followed by restaging studies and immune assessments at day +100. At day 100, after immunizations and restaging, patients will start Revlamid® (Lenalidomide) maintenance therapy followed by 2 additional MAGE-A3 and PCV immunizations at days 120 and 150.
  Interventions: Biological: Prevnar- Pneumococcal Conjugate Vaccine (PCV); Other: Activated/costimulated autologous T-cell; Drug: Revlamid® (Lenalidomide); Biological: MAGE-A3/GM-GSF, Hiltonol® (Poly-ICLC)

INTERVENTIONS:
Biological: Prevnar- Pneumococcal Conjugate Vaccine (PCV) — After study enrollment, patients will receive Prevnar- Pneumococcal Conjugate Vaccine (PCV). At Day #14, Day #42, and Day #90, Day #120 and Day #150, patients will receive a booster immunization with Prevnar- Pneumococcal Conjugate Vaccine (PCV).
Other: Activated/costimulated autologous T-cell — For all patients, the cells will be expanded ex vivo for up to 12 days and then prepared for infusion ~day 2 post-transplant. The target number of costimulated T-cells for infusion will be ~ 5 x 10e10 T-cells total in 100-500 mL total volume.
Drug: Revlamid® (Lenalidomide) — At about day 100 post-transplant, after completion of post-transplant immunological assessments and myeloma restaging studies, patients will be eligible to receive low-dose Revlamid® (Lenalidomide) 10 mg/day for maintenance therapy (10 mg/day) until progression of myeloma or development of intolerance.
Biological: MAGE-A3/GM-GSF, Hiltonol® (Poly-ICLC) — After study enrollment, patients will receive both MAGE-A3/GM-CSF [+ coinjection of 2mg of Hiltonol®(Poly-ICLC)]. At Day #14, Day #42, Day #90, Day #120 and Day #150 patients will receive an additional immunization with MAGE-A3/GM-GSF, Hiltonol® (Poly-ICLC).

SUMMARY:
One purpose of this study is to find out if a new combination of immune system treatments (MAGE-A3 vaccine plus activated T-cells) will allow the body to build up protection ("immunity") against the myeloma cells. A second purpose is to find out how well this combination of immune system treatments is able to control the myeloma.

DETAILED DESCRIPTION:
Autologous stem cell transplant (ASCT) can lead to a complete or partial disappearance of the myeloma in about 2 out of 3 patients. However, an ASCT only sometimes leads to a cure of the myeloma. In about half the patients the myeloma comes back after about 1-2 years. In about 90% of patients it comes back by about 10 years after transplant.

One possible way to improve upon the results of ASCT for myeloma is to help the body's defense or immune system recover faster after transplant. Another way is to teach the body's immune system to fight against the myeloma cells.

In two earlier research studies which included more than 100 patients, certain types of immune cells called "T cells" or "T lymphocytes" were taken out of a patient's body using a procedure called "apheresis". These cells were then grown up in the lab. After the transplant, these T cells were put back into the patients. The replaced T cells helped the patients'immune systems to recover faster after the transplant. In addition, when the T cells were given back to patients they also received a vaccination. The vaccination or injection was for a certain type of pneumonia germ called "pneumococcus". We found that most patients built up protection against this pneumonia-causing germ. In another study, we used a possible myeloma cancer vaccine. However, we found that less than half the patients responded to this vaccine.

In this new study, we want to test a different type of myeloma cancer vaccine. This different cancer vaccine is based on a protein called MAGE-A3. The MAGE-A3 protein is found in about 50% of cases of myeloma. This vaccine consists of small pieces of protein (called "peptides") which come from the MAGE-A3 protein. In order to help the immune system respond better we will add two new steps. First we will add an immune system stimulant called "Hiltonol®" to each vaccination. Hiltonol® is a chemical substance that turns on several parts of the immune system. It may make the immune system better able to respond to the vaccine. It has been tested in several hundred patients and has been used with about a dozen different types of cancer and germ vaccines. Second, starting about 100 days after the transplant procedure, patients will get a medicine called Lenalidomide. Lenalidomide is already approved by the Food and Drug Administration (FDA) for treatment of myeloma. In this study, we want to know whether Lenalidomide could help to improve the body's ability to respond to the vaccinations and help to treat the myeloma itself.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Patients must be registered with the Sponsor's Monitor
* Patients must have a diagnosis of myeloma
* Patients must meet one of the following criteria:

  1. Myeloma has relapsed, progressed, or failed to respond after at least one prior course of therapy (consisting of at least 2 treatment cycles or months of therapy).
  2. Myeloma has responded partially to initial therapy but a complete response (immunofixation negative and normal serum free light chain studies)has NOT developed after a minimum of 3 cycles or months of initial therapy.
  3. Myeloma has high-risk features as defined by the presence of one or more cytogenetic abnormalities known to confer a poor outcome even after standard autotransplants:complex karyotype (> or = to 3 abnormalities),t(4;14),t(14;16),del (17)(p13.1),and/or chromosome 13 abnormalities.
* Patients must have measurable disease on study entry
* Patients must be between ages 18-80 (inclusive).
* Patients should have adequate vital organ function as defined by the protocol.
* ECOG performance status 0-2 (unless due solely to bone pain)
* Prior to Lenalidomide maintenance phase, all study participants must be registered into the mandatory RevAssist® program, and be willing and able to comply with the requirements of RevAssist®.
* Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test as per the protocol
* Lenalidomide treatment phase: able to take aspirin (81 or 325 mg) daily as prophylactic anticoagulation (patients intolerant to ASA may use warfarin or low molecular weight heparin).

Exclusion Criteria:

* Pregnant or nursing females
* HIV or HTLV-1/2 seropositivity
* Known history of myelodysplasia
* Known history of chronic active hepatitis or liver cirrhosis (if suspected by laboratory studies, should be confirmed by liver biopsy).
* Active Hepatitis B (as defined by + Hepatitis B surface antigen); + Hepatitis C virus (HCV) antibody is NOT an exclusion
* Prior autotransplant or allogeneic transplant
* More than 4 distinct, prior courses of therapy for myeloma
* History of severe autoimmune disease requiring steroids or other immunosuppressive treatments.
* Active immune-mediated diseases including:connective tissue diseases, uveitis,sarcoidosis,inflammatory bowel disease, multiple sclerosis.
* Evidence or history of other significant cardiac,hepatic,renal, ophthalmologic,psychiatric,or gastrointestinal disease which would likely increase the risks of participating in the study
* Active bacterial, viral or fungal infections.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2011-05-10 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Rapoport, M.D., Study Chair — University of Maryland Greenebaum Cancer Center; Ed Stadtmauer, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (2):
- United States (2):
  - University of Maryland Greenebaum Cancer Center, Baltimore, Maryland
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Rapoport AP, Aqui NA, Stadtmauer EA, Vogl DT, Xu YY, Kalos M, Cai L, Fang HB, Weiss BM, Badros A, Yanovich S, Akpek G, Tsao P, Cross A, Mann D, Philip S, Kerr N, Brennan A, Zheng Z, Ruehle K, Milliron T, Strome SE, Salazar AM, Levine BL, June CH. Combination immunotherapy after ASCT for multiple myeloma using MAGE-A3/Poly-ICLC immunizations followed by adoptive transfer of vaccine-primed and costimulated autologous T cells. Clin Cancer Res. 2014 Mar 1;20(5):1355-65. doi: 10.1158/1078-0432.CCR-13-2817. Epub 2014 Feb 11. PMID 24520093

RESULTS

PARTICIPANT FLOW:
Groups:
- MAGE A-3, GM-CSF, Hiltonol®, T Cells, Lenalidomide,: MAGE-A3, GM-CSF, Hiltonol® (Poly-ICLC), PCV vaccine prior to apheresis.
  Stem cell mobilization. High-dose melphalan, then hematopoietic stem cells on Day 0.
  Day 2 Activated/costimulated autologous T cells.
  Days 14, 42 and 90 MAGE-A3, Hiltonol® and PVC.
  Day 100 start Lenalidomide.
  Day 120 and 150 MAGE-A3 and PVC.
Period: Enrollment
Arm/Group | MAGE A-3, GM-CSF, Hiltonol®, T Cells, Lenalidomide,
Started | 28
Completed | 27 (One subject failed to meet screening criteria for the trial.)
Not Completed | 1
Period: Pre Transplant Vaccinations
Arm/Group | MAGE A-3, GM-CSF, Hiltonol®, T Cells, Lenalidomide,
Started | 27
Pre Transplant Vaccinations 1-3 (MAGE-A3, GM-CSF, Hiltonol®, PCV vaccine ~10 days before apheresis.) | 27
Completed | 27
Not Completed | 0
Period: Activated/Costimulated Autologous T Cell
Arm/Group | MAGE A-3, GM-CSF, Hiltonol®, T Cells, Lenalidomide,
Started | 27
Completed | 27
Not Completed | 0
Period: MAGE-A3, Hiltonol®, PVC After T Cells
Arm/Group | MAGE A-3, GM-CSF, Hiltonol®, T Cells, Lenalidomide,
Started (On study Days 14, 42 and 90 study participants will receive MAGE-A3, Hiltonol® and PVC vaccine.) | 27
Completed | 26
Not Completed | 1
Not completed — Off Study due to Disease Progression | 1
Period: Start Lenalidomide
Arm/Group | MAGE A-3, GM-CSF, Hiltonol®, T Cells, Lenalidomide,
Started | 26
Completed | 26
Not Completed | 0
Period: Maintenance: MAGE-A3, PVC After T Cells
Arm/Group | MAGE A-3, GM-CSF, Hiltonol®, T Cells, Lenalidomide,
Started | 26
Completed | 26
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Prevnar, T Cells, Lenalidomide, MAGE A-3: MAGE-A3, GM-CSF, Hiltonol® (Poly-ICLC), PCV vaccine prior to apheresis.
  Stem cell mobilization. High-dose melphalan, then hematopoietic stem cells on Day 0.
  Day 2 Activated/costimulated autologous T cells.
  Days 14, 42 and 90 MAGE-A3, Hiltonol® and PVC.
  Day 100 start Lenalidomide.
  Day 120 and 150 MAGE-A3 and PVC.
Arm/Group | Prevnar, T Cells, Lenalidomide, MAGE A-3
Number analyzed (Participants) | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 5
Age, Continuous [Mean (Full Range); unit: years] | 52.48 [42 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 18
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 27

OUTCOME MEASURES:

1. Primary Outcome: Primary Myeloma Endpoint
Description: To determine whether lenalidomide maintenance plus the late booster immunizations leads to improved myeloma clinical responses between day 180 and day 100 post-transplant.
Time Frame: Between day 100 and 180 post transplant
Population: Subjects that reached D100 and D180
Measure: Count of Participants; unit: Participants
Groups:
- Prevnar, T Cells, Lenalidomide, MAGE A-3: All patients will receive a priming immunization with a MAGE-A3/GM-CSF vaccine with adjuvant Hiltonol® (Poly-ICLC) along with the pneumococcal conjugate vaccine/PCV control vaccine about 10 days before a steady-state mononuclear cell apheresis. Patients will then undergo hematopoietic stem cell mobilization. All patients will receive high-dose melphalan followed by hematopoietic stem cells on day 0.
Arm/Group | Prevnar, T Cells, Lenalidomide, MAGE A-3
Number analyzed (Participants) | 26
Participants
  Subjects in CR D100 and D180 | 4
  Subjects in sCR D100 and 180 | 1
  Subjects in VGPR D100 and D180 | 1
  Subjects in PR D100 and D180 | 5
  Subjects with SD at D+100 and 180 | 3
  Subjects with improved response at D100 and D180 | 6
  Subjects with poorer response at D100 and D180 | 4
  Subjects with no disease response reported | 2

ADVERSE EVENTS:
Time Frame: Adverse event reporting begins at the time of T-cell harvest and continues until day 180 post infusion.
Arm/Group | Prevnar, T Cells, Lenalidomide, MAGE A-3
All-Cause Mortality (participants affected / at risk) | 0/27
Serious Adverse Events (participants affected / at risk) | 9/27
Other Adverse Events (participants affected / at risk) | 27/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prevnar, T Cells, Lenalidomide, MAGE A-3 (N=27)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Coughing/shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Fever (General disorders) | 2 (2)
Flu like symptoms (General disorders) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Hypothermia (General disorders) | 1 (1)
Influenza B (Infections and infestations) | 1 (1)
Infusion site Extravasation (General disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Nausea/Vomiting (Gastrointestinal disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 3 (3)
Platelet count decreased (Investigations) | 2 (2)
Pneumonia (Infections and infestations) | 4 (5)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Skin Indurations w/erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Sterile abscess w/drainage (Infections and infestations) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prevnar, T Cells, Lenalidomide, MAGE A-3 (N=27)
Anorexia (Metabolism and nutrition disorders) | 9 (14)
Chills (General disorders) | 5 (7)
Diarrhea (Gastrointestinal disorders) | 4 (5)
Fatigue (General disorders) | 7 (7)
Fever (General disorders) | 10 (16)
Flu-like symptoms (Infections and infestations) | 2 (3)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Headache (Nervous system disorders) | 8 (10)
Increased eosinophil (Blood and lymphatic system disorders) | 2 (3)
Induration (Skin and subcutaneous tissue disorders) | 3 (5)
Induration - thigh (Skin and subcutaneous tissue disorders) | 2 (2)
Induration at injection site (Skin and subcutaneous tissue disorders) | 7 (14)
Induration/Swelling (Skin and subcutaneous tissue disorders) | 4 (7)
Injection site reaction (General disorders) | 8 (36)
Loss of energy (Nervous system disorders) | 8 (13)
Muscle aches (Musculoskeletal and connective tissue disorders) | 11 (17)
Nausea (Gastrointestinal disorders) | 5 (6)
Neutrophil count decreased (Investigations) | 2 (2)
Pain at injection site (Gastrointestinal disorders) | 16 (40)
Pruritis (Skin and subcutaneous tissue disorders) | 2 (3)
Rash (Skin and subcutaneous tissue disorders) | 3 (3)
Rash - lower extremity (Skin and subcutaneous tissue disorders) | 2 (2)
Swelling at injection site (General disorders) | 2 (2)
Swelling/Induration (Musculoskeletal and connective tissue disorders) | 7 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No